CLINICAL TRIAL: NCT02259036
Title: Using Smartphones to Enhance the Treatment of Childhood Anxiety
Acronym: Smart-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Silk, PhD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH102666; 1R34MH102666-01A1 (NIH)
Record Dates: First submitted 2014-09-24; First posted 2014-10-08 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Anxiety
Keywords: child anxiety; worries; fears; talk therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SmartCAT Enhanced Treatment (Other): Cognitive Behavioral Therapy enhanced with an ecological momentary treatment enhancement smartphone app called SmartCAT.
  Interventions: Other: Ecological Momentary Treatment Enhancement

INTERVENTIONS:
Other: Ecological Momentary Treatment Enhancement — Participants will be given a pre-programmed smartphone on which they will enter their responses to a series of questions about moods and daily experiences using an app developed for this study. The child will receive an electronic notification message once per day and will be prompted through a series of questions about what he/she is doing, who he/she is with, how he/she is feeling, worries or stressful events, and how he/she coped with these events. It should take the child approximately 5 minutes each time to complete the questions. Participant data will be sent to study therapists to be reviewed weekly. The therapist will integrate this information into treatment and provide customized feedback to the patient.

SUMMARY:
The primary goal of this research study is to develop an interactive smartphone app that could be used to increase the effectiveness of talk therapy such as cognitive behavioral therapy (CBT) for child anxiety.

DETAILED DESCRIPTION:
Boys and girls between the ages of 9-14 who have anxiety and a parent or caregiver are being asked to participate in this study. Interested participants who contact the study will be asked to undergo a brief phone pre-screen to determine initial eligibility.

After completing a phone pre-screen, potential participants for the Phase 2 trial will be invited to the lab to complete a clinical intake interview. Clinical information will be obtained from parent and child by a trained research staff member. The research staff member will have specific training to a high degree of reliability in conducting the diagnostic interviews relevant to this research study.

Participants that meet study criteria based on the clinical information obtained at the first study visit will be invited to begin a course of Cognitive Behavior Therapy (CBT), an empirically validated talk therapy commonly used to treat children with anxiety. Children will receive individual treatment using the Brief Coping Cat Manual. The Coping Cat program (Kendall 1994) is an empirically supported child-focused CBT treatment for children with anxiety disorders. Throughout the program, children are encouraged to practice techniques learned during therapy sessions through homework or "Show-That-I-Can" (STIC) tasks. Parents attend weekly check-ins and two parent-only sessions. STIC tasks will consist of specific SmartCAT modules in the smartphone app as assigned at the end of each session. Participants might be asked to interact with other children and adolescents or study staff as well as leave the therapy building. This is to allow participants to become more comfortable in situations that make them feel anxious by gradually exposing them to the specific situation. Parents are not treated as co-clients, but are considered consultants to the child's treatment and are asked to provide some collaboration and assistance in exposure planning and homework.

Treatment will be delivered by Masters-level therapists who will have completed training in CBT. They will attend a weekly supervision session with Dr. Silk, with consultation from Dr. Kendall on difficult cases via videoconference. All sessions will be videotaped.

SMARTPHONE PROTOCOL:

Prior to the first therapy session, the child and a parent will be trained how to use the SmartCAT app. Youth will be provided with an Android smartphone for the duration of the study. If the child already has an Android phone, the app will be installed on the participant's phone in order to decrease participant burden of carrying an additional phone.

Participants will be given a study-provided, pre-programmed smartphone on which they will enter their responses to a series of questions about moods and daily experiences using an app developed for this study. The child will receive an electronic notification message once per day and will be prompted through a series of questions about what he/she is doing, who he/she is with, how he/she is feeling, worries or stressful events, and how he/she coped with these events. It should take the child approximately 5 minutes each time to complete the questions. The child will only be prompted to answer these questions outside of school hours and on weekends. Participant data will be securely sent to study therapists via a clinician portal connected to the app to be reviewed weekly. The therapists may then integrate this information into treatment and provide customized feedback to the patient.

Parents will be asked to complete an online diary to keep track of what skills their child uses during the week. After completion of the initial screening visit, parents are asked to complete the Skills Use Diary daily for seven days. After this seven day period, they will be asked to complete a diary entry twice per week throughout 8 weeks of treatment, totaling 30 entries. At the end of treatment, subjects will again be asked to complete the diary daily for another seven days. Participants will receive links to the online diary and instructions for completion via email (see references and other attachments for the email script). Diaries should take no longer than 10 min per day to complete. The data will be encrypted and stored securely through the online survey system Qualtrics.

POST-TREATMENT and 2-MONTH FOLLOW-UP:

All clinical, skill acquisition, and skill utilization measures (including the parent 7 day diary) will be repeated at post-treatment (approximately 10 weeks) and 2 month follow-up We will use Qualtrics, a secure internet data collection system, for administering diaries and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 40 children of either sex ages 9 years, 0 months to 14 years, 11 months with DSM-IV diagnosis of Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SAD), and/or Social Phobia (SP) as identified by the Kiddie Schedule of Affective Disorders.

The primary caregiver is defined as the person who has the most responsibility for taking care of the child. While this is typically the mother, it can be the father, an adoptive parent or other legal guardian. The primary caregiver must be a legal guardian of the child.

Exclusion Criteria:

1. Requires current ongoing treatment with psychoactive medications other than stimulants.
2. Acutely suicidal or at risk for harm to self or others.
3. Neuromuscular or neurological disorder.
4. Reading level below 80 on the Wide Range Achievement Test-4 (WRAT-4)
5. Medical illnesses or medications taken for an illness as determined by study physicians that would affect study adherence, and subject's emotional state.
6. Current comorbid diagnosis of: primary major depressive disorder (MDD) (subjects who have primary GAD with co-morbid MDD that is secondary in terms of course and functional impact are not excluded), obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), conduct disorder, substance abuse or dependence, and ADHD combined type or predominantly hyperactive-impulsive type.
7. Lifetime diagnosis of autism spectrum disorder, bipolar disorder, psychotic depression, schizophrenia, or schizoaffective disorder.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
PARS Treatment response | 10 weeks
  Anxiety severity will be rated by an IE on the Pediatric Anxiety Rating Scale (PARS) (RUPP Study Group, 2002). A total score was computed by summing six items assessing anxiety severity, frequency, distress, avoidance, and interference during the previous week. Treatment response will be defined as a 35% reduction in PARS from pre- to post-treatment.

SECONDARY OUTCOMES:
Absence of diagnosis on K-SADS | 10 weeks
  Recovery will be defined as an absence of DSM 5 diagnosis of Separation Anxiety, Social Anxiety, and Generalized Anxiety Disorder on the K-SADS interview.

OTHER OUTCOMES:
child report of anxiety | 10 weeks
  child report of anxiety severity on the Screen for Childhood Anxiety Related Emotional Disorders (SCARED).
parent report of anxiety | 10 weeks
  parent report of anxiety severity on the Screen for Childhood Anxiety Related Emotional Disorders (SCARED).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Silk, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Dept. of Psychology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achenbach, T. M. (1991). Manual for the Child Behavior Checklist/4-18 and 1991 Profile. Burlington: University of Vermont, Department of Psychiatry.
- [Background] Angold, A., Costello, E. J., Messer, S. C., Pickles, A., Winder, F., & Silver, D. (1995). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents. Interenational Journal of Methods in Psychiatric Research, 5, 237-249.
- [Background] Birmaher, B., Khetarpal, S., Cully, M., Brent, D. A., & McKenzie, S. (2003). Screen for Child Anxiety Related Disorders (SCARED)--Parent form and child form (8 years and older). In L. VandeCreek (Ed.), Ellis Human Development Institute. (pp. 99-104). Sarasota, FL: Professional Resource Press/Professional Resource Exchange, Inc.
- [Background] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Background] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Background] Connor-Smith JK, Compas BE, Wadsworth ME, Thomsen AH, Saltzman H. Responses to stress in adolescence: measurement of coping and involuntary stress responses. J Consult Clin Psychol. 2000 Dec;68(6):976-92. PMID 11142550
- [Background] Constantino, J. N. (2002). The Social Responsiveness Scale, Los Angeles: Western Psychological Services.
- [Background] Guy W (1976): The clinical global impression scale. The ECDEU Assessment Manual for Psychopharmacology-Revised Rockville, MD U.S. Department of Health, Education, and Welfare Public Health Service, Alcohol, Drug Abuse, Mental Health Administration, NIMH Psychopharmacology Research Branch, Division of Extramural Research.
- [Background] Harter, S. (1988). Manual for the Self-perception Profile for Adolescents Denver, CO: University of Denver.
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kendall PC. Treating anxiety disorders in children: results of a randomized clinical trial. J Consult Clin Psychol. 1994 Feb;62(1):100-10. doi: 10.1037//0022-006x.62.1.100. PMID 8034812
- [Background] Langley AK, Bergman RL, McCracken J, Piacentini JC. Impairment in childhood anxiety disorders: preliminary examination of the child anxiety impact scale-parent version. J Child Adolesc Psychopharmacol. 2004 Spring;14(1):105-14. doi: 10.1089/104454604773840544. PMID 15142397
- [Background] Reynolds S, Wilson C, Austin J, Hooper L. Effects of psychotherapy for anxiety in children and adolescents: a meta-analytic review. Clin Psychol Rev. 2012 Jun;32(4):251-62. doi: 10.1016/j.cpr.2012.01.005. Epub 2012 Feb 13. PMID 22459788
- [Background] Pine DS, Cohen P, Gurley D, Brook J, Ma Y. The risk for early-adulthood anxiety and depressive disorders in adolescents with anxiety and depressive disorders. Arch Gen Psychiatry. 1998 Jan;55(1):56-64. doi: 10.1001/archpsyc.55.1.56. PMID 9435761
- [Background] Ronan, K. R., Kendall, P. C., & Rowe, M. (1994). Negative affectivity in children: Development and validation of a self-statement questionnaire. Cognitive Therapy and Research, 18(6), 509-528.
- [Background] The Pediatric Anxiety Rating Scale (PARS): development and psychometric properties. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1061-9. doi: 10.1097/00004583-200209000-00006. PMID 12218427
- [Background] Silk JS, Dahl RE, Ryan ND, Forbes EE, Axelson DA, Birmaher B, Siegle GJ. Pupillary reactivity to emotional information in child and adolescent depression: links to clinical and ecological measures. Am J Psychiatry. 2007 Dec;164(12):1873-80. doi: 10.1176/appi.ajp.2007.06111816. PMID 18056243
- [Background] Silk JS, Forbes EE, Whalen DJ, Jakubcak JL, Thompson WK, Ryan ND, Axelson DA, Birmaher B, Dahl RE. Daily emotional dynamics in depressed youth: a cell phone ecological momentary assessment study. J Exp Child Psychol. 2011 Oct;110(2):241-57. doi: 10.1016/j.jecp.2010.10.007. Epub 2010 Nov 26. PMID 21112595
- [Background] Silk JS, Steinberg L, Morris AS. Adolescents' emotion regulation in daily life: links to depressive symptoms and problem behavior. Child Dev. 2003 Nov-Dec;74(6):1869-80. doi: 10.1046/j.1467-8624.2003.00643.x. PMID 14669901
- [Background] Zeman, J., Shipman, K., & Penza Clyve, S. (2001). Development and initial validation of the Children's Sadness Management Scale. Journal of Nonverbal Behavior, 25(3), 187-205.
- [Background] Ziegert DI, Kistner JA. Response styles theory: downward extension to children. J Clin Child Adolesc Psychol. 2002 Sep;31(3):325-34. doi: 10.1207/S15374424JCCP3103_04. PMID 12149970
- [Derived] McCormack CC, Mennies RJ, Silk JS, Stone LB. How anxious is too anxious? State and trait physiological arousal predict anxious youth's treatment response to brief cognitive behavioral therapy. BMC Psychol. 2020 May 12;8(1):48. doi: 10.1186/s40359-020-00415-3. PMID 32398128